CLINICAL TRIAL: NCT05394714
Title: A Dose-Escalating Phase I Study to Determine the Safety, and Maximum Tolerated Dose/ Maximum Feasible Dose of Autologous ex Vivo Expanded and Activated NK Cell, Magicell-NK, Infusion for Colon Cancer Post Resection
Brief Title: A Phase I, Autologous ex Vivo Expanded and Activated NK Cell, Magicell-NK, Infusion for Colon Cancer Post Resection Study
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Medigen Biotechnology Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CT-NK-11
Record Dates: First submitted 2022-05-11; First posted 2022-05-27 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Colon Cancer Stage I
MeSH Terms: conditions — Colonic Neoplasms | interventions — Saline Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Magicell-NK (Experimental): Magicell-NK Cohort 1: 2 x 10^8 cells x 6 infusions Cohort 2: 6 x 10^8 cells x 6 infusions Cohort 3: 12~18 x 10^8 cells x 6 infusions
  Interventions: Biological: Magicell-NK contains NK cells suspended in 100 mL normal saline

INTERVENTIONS:
Biological: Magicell-NK contains NK cells suspended in 100 mL normal saline — Eligible subjects will be assigned into one of the three dose escalating cohorts (3+3 subjects/cohort) according to the time sequence enrolled

SUMMARY:
This is a Phase I, open-label study to explore the safety profile and to find the maximum tolerated dose (MTD) or maximum feasible dose (MFD) of Magicell-NK in subjects diagnosed with stage I or stage IIa colon cancer post resection from a single site in Taiwan.

During this study, 3 dose levels of Magicell-NK will be tested with a 3+3 design to determine the MTD/MFD: Cohort 1, low dose (2×10^8 cells), Cohort 2, middle dose (6×10^8 cells), and Cohort 3, high dose (12~18 ×10^8 cells).

ELIGIBILITY:
Inclusion Criteria:

1. A dated and signed informed consent
2. Either gender and aged over 20 years old (inclusive) at date of consent
3. With histologically confirmed stage I or stage IIa colon cancer
4. Received curative colon resection within 4~8 weeks prior to the screening visit and does not need adjuvant chemotherapy or radiotherapy
5. With no ≥ grade 3 postoperative complications or has been recovered and is suitable for study enrollment according to the investigator's judgment
6. With adequate hematology function:

   * Absolute neutrophil count (ANC) ≥ 1,500 cells/μL
   * Total white blood cell (WBC) ≥ 3,000 cells/μL
   * Platelets ≥ 100,000 counts/μL
   * Hemoglobin ≥ 9 g/dL
7. With adequate hepatic and renal function:

   * Serum creatinine ≤ 1.5 × Upper Limit of Normal (ULN)
   * Total bilirubin (TB) ≤ 1.5 × ULN
   * ALT and AST ≤ 2.5 × ULN
   * Alkaline phosphatase (ALP) ≤ 5X ULN
8. Negative response in HIV and syphilis test
9. Subject with childbearing potential must agree to abstain from intercourse or use highly effective contraceptives from when signing informed consent to the Final/ET Visit.
10. Performance status (ECOG) < 2
11. Patients agree to be in compliant to clinical protocol planned treatment plan

Exclusion Criteria:

1. Received any other investigational, anti-neoplastic medication (except squamous cell carcinoma, basal cell carcinoma, or carcinoma in situ of the skin, curatively treated with cryosurgery or surgical excision only), or immune cell therapy within 28 days prior to Day 1.
2. Currently under immunosuppressive or systemic steroid treatment with equivalent dosage higher than prednisolone 30 mg/day for more than 7 days within 14 days prior to Day 1
3. With known tumor metastasis or coexisting malignant disease
4. With ongoing acute diseases, or within the past 2 years having serious medical conditions (e.g. concomitant illness) such as cardiovascular (e.g. New York Heart Association grade III or IV), hepatic (e.g. Child-Pugh Class C), psychiatric condition (e.g. alcoholism, drug abuse), medical history, physical findings, or laboratory abnormality that, judged by the investigator, could interfere with the results of the trial or adversely affect the safety of the subject
5. Known hypersensitivity to aminoglycoside or bacitracin (e.g. Streptomycin, Gentamicin)
6. Known hypersensitivity to any of the components of Magicell-NK, including human serum albumin
7. Female subject who is lactating or has positive urine pregnancy test at screening

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2022-03-10 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Serious Adverse Events (SAEs) and Treatment Emergent Adverse Events (TEAEs) | Up to 60 weeks
  Number of participants with serious adverse events and treatment emergent adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0) to assess tolerability of Magicell-NK treatment. Evaluation of side effects conducted during the study period. A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Number of Participants With at Least One Dose Limiting Toxicity | Within 14-day observation of the first treatment. up to 60 weeks
  Dose Limiting Toxicity (DLT) as defined by the Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0 as treatment-related any greater or equal to Grade 4 adverse event of hematologic toxicity, or any greater or equal to Grade 3 adverse event of non-hematologic toxicity during Visit 3~ visit 10. With the exception of (1) fever grade 3 or grade 4 which is controllable by antihistamine and resolves to grade 2 or less within 48 hours, (2) hypersensitivity reactions occurring within 2 hours of infusion finished (related to cell infusion) that are reversible to a grade 2 or less within 48 hours with standard therapy, (3) grade 3 electrolyte imbalance or dehydration that resolves to grade 1 or less within 48 hours, (4) grade 3 nausea, vomiting, or diarrhea which is controllable by standard medication that resolves to grade 1 or less within 48 hours, (5) fatigue which resolves to grade 1 or less within 7 days.
Maximum Tolerated Dose (MTD) and Recommended Phase II Dose (RP2D) | 3 weeks from start of treatment, up to 60 weeks
  MTD is defined as the highest dose level at which ≤ 1/6 of subjects experiences DLT during Visit 3~10, when at least 6 patients are treated at that dose and are evaluable for toxicity. Dose escalations proceeded according to a standard 3+3 design. Maximum tolerated dose (MTD) and recommended phase II dose (RP2D) of therapy was determined by monitoring dose-limiting toxicity and adverse events in the dosing cohorts

SECONDARY OUTCOMES:
Disease free survival (DFS) | Up to 60 weeks
  The time from the date of the first Magicell-NK infusion to the date of the first disease-free survival event (recurrence, second primary colon cancer or death from any cause).
Changes in Frequency and Duration of ctDNA | Up to 60 weeks
  Number of participants experiencing ctDNA seroconversion (i.e. ctDNA+ that become ctDNA-) after any Magicell-NK regimen remaining disease free. Change in values will be tabulated descriptively by visit with 95% two-sided confidence interval.
Changes in Frequency and Duration of Circulating Tumor Count (CTC) and Programmed Death-Ligand 1 Circulating Tumor Count (PD-L1+ CTC) counts | Up to 60 weeks
  Determine the effect of Magicell-NK on reducing CTC and PD-L1+ CTC of whole blood in colon cancer with elevated baseline CTC count and PD-L1+ CTC to identify the least effective dose that clears CTCs and PD-L1+ CTC. Baseline count of CTC and PD-L1+ CTC will be recorded prior to before Magicell-NK therapy in a whole blood sample. Count of CTC and PD-L1+ CTC will be measured at 1 week (post treatment evaluation visit), and 10-12 weeks (follow up visits) after Magicell-NK therapy in a whole blood sample. These values will be compared.
Changes in Biomarkers (CEA and CA19-9) | Up to 60 weeks
  Determine the effect of Magicell-NK on CEA and CA 19-9 in colon cancer with elevated baseline CEA and CA 19-9 to identify the least effective dose that clears CEA and CA 19-9. Baseline count of CEA and CA 19-9 will be recorded prior to before Magicell-NK therapy. Count of CEA and CA 19-9 will be measured at 1 week (post treatment evaluation visit), and 10-12 weeks (follow up visits) after Magicell-NK therapy. These values will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Stanley Chang, PhD, Study Chair — Medigen Biotechnology Corporation
Locations (1):
- Chang Gung Memorial Hospital, Linkou, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No